CLINICAL TRIAL: NCT05705765
Title: Effects on Balance in the Young Adult of Suspension Exercise vs. Exercise on Unstable Surfaces: a Quasi-randomized Clinical Trial
Brief Title: Effects on Balance of Suspension Exercise vs. Exercise on Unstable Surfaces
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, David Hernández-Guillén, Assistant professor, PT, PhD, University of Valencia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SUS_VS_INEST
Record Dates: First submitted 2023-01-20; First posted 2023-01-31 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Balance Training; Instability
Keywords: Suspension training; Instability training; Balance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suspension (Experimental): Exercise with suspension devices.
  Interventions: Other: Suspension training
- Balance (Active Comparator): Exercise over instability surfaces.
  Interventions: Other: Instability training

INTERVENTIONS:
Other: Suspension training — Training with suspension devices. 12 sessions of 40-45 min in four weeks.
  Arms: Suspension
Other: Instability training — Training on unstable surfaces. 12 sessions of 40-45 min in four weeks.
  Arms: Balance

SUMMARY:
Most human movements are executed while in a state of postural instability. For this reason, instability training is a highly-specific method that is intended to improve balance and postural control. This research aimed to determine the effect of instability training on the balance of individuals with similar baseline abilities, who initiated training within different stability conditions. Research question: Does different type of instability training determine improvements in balance?

ELIGIBILITY:
Inclusion Criteria:

* University students aged 18-35 years.

Exclusion Criteria:

* Muscle skeletal injury in the preceding 6 months.
* Athletes from any field.
* Those with known blance disorders (e.g. vertigo and central or vestibular disorder).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Y Balance Test | 0 week
  The Y Balance Test is a portion of the Functional Movement Systems screen used to evaluate dynamic balance and functional symmetry in order to determine a person's risk for injury or return to sport readiness. Procedure: The starting position is standing on one leg at the stance plate with the toes of the foot at the red line, and the other leg touching down lightly just behind the plate. The non-stance foot is reached out in the desired direction, pushing the reach indicator as far as they can while maintaining balance. The higher the value, the better the balance.
Y Balance Test | 5 week
  The Y Balance Test is a portion of the Functional Movement Systems screen used to evaluate dynamic balance and functional symmetry in order to determine a person's risk for injury or return to sport readiness. Procedure: The starting position is standing on one leg at the stance plate with the toes of the foot at the red line, and the other leg touching down lightly just behind the plate. The non-stance foot is reached out in the desired direction, pushing the reach indicator as far as they can while maintaining balance. The higher the value, the better the balance.

SECONDARY OUTCOMES:
Emery Test | 0 week, 5 week.
  Monopodal balance on an unstable base. The time that is held with closed eyes is counted before losing balance. The longer it is held, the better the balance is considered.
Romberg Test | 0 week, 5 week.
  Bipodal balance on pressure platform. They hold on for 30 seconds with their eyes open. This test gives data on the area and speed of displacement of the center of gravity. The lower the values, the better the balance.
Sidewide Test | 0 week, 5 week
  The participant will perform side jumps over a 25 cm wide board. The number of jumps you make will be counted. The higher the number of jumps, the agility will be considered to be better.

CONTACTS AND LOCATIONS:
Overall Officials: David Hernández-Guillén, PT, PhD, Principal Investigator — University of Valencia
Locations (1):
- Faculty of Physiotherapy of the University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No